CLINICAL TRIAL: NCT00274664
Title: Randomised Occlusion Treatment of Amblyopia Study (ROTAS): Trial of Maximal Vs Substantial Doses of Occlusion to Evaluate Visual Outcome for Children With Amblyopia
Brief Title: Patching for Lazy Eye: Trial to Evaluate Daily Patching Amounts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: Imperial College London (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROTAS-091206; Fight for Sight: 20500
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2006-01-11 (Estimated); Status verified 2005-12

CONDITIONS: Amblyopia
Keywords: Amblyopia; Occlusion dose monitoring; Refractive adaptation; Dose-response
MeSH Terms: conditions — Amblyopia

INTERVENTIONS:
Device: 6 hours occlusion by patching
Device: 12 hours occlusion by patching

SUMMARY:
Amblyopia ('lazy eye') is the commonest visual disorder of childhood and is caused by an interruption to visual development. Occlusion of the better eye by patching is the mainstay of treatment, so forcing use, of the affected eye. We have little understanding of how much treatment is required for improvement, so occlusion may continue for many months. This is both demanding for the child and family as a whole. Treatment outcome is frequently unsatisfactory. Compliance is often poor, thus we do not know precisely how much treatment the child actually receives or how much is required.

To overcome this, we have designed an instrument that permits us to measure occlusion: an occlusion dose monitor (ODM) which provides an objective record of how much occlusion a child actually receives. Recently we have observed that 75% of improvement induced by occlusion occurs in the first four weeks of treatment. In this study we explore the possibility that by intensive treatment the period of amblyopia therapy can be shortened - i.e. treatment will be more efficient, more effective, and more 'family-friendly'. The study hypothesis is that 12 hours/day of patching is more effective than 6 hours/day.

DETAILED DESCRIPTION:
The identification and subsequent management of amblyopia are major consumers of health service resource, and within the hospital sector account for around 80-90% of visits to the children's eye service. Occlusion of the better eye is the mainstay of treatment and because we have little understanding of the dose-response relationship this may continue for many months and sometimes for many hundreds of hours. This is demanding for the child and family as a whole and yet the outcome is frequently unsatisfactory. Currently, there is no reliable data on the kinetics of visual improvement, so occlusion tends to be prescribed on an ad hoc basis. Recent pilot research has shown that 75% of the treatment-generated improvement occurs within the first 4 weeks when 6 hours/day occlusion is prescribed.

In this study we explore the possibility that by intensive treatment the period of amblyopia therapy can be shortened - i.e. made both more efficient and hopefully more effective. The purpose of the present study, the Randomized Occlusion Treatment of Amblyopia Study (ROTAS), is to compare two frequently employed patching regimens: 'substantial' (6 hrs/day) against 'maximal' (12 hrs/day) patching. Our experimental design incorporates objective occlusion monitoring and is able to discriminate the beneficial effect of refractive correction from that of occlusion. The study comprises three phases: 'baseline', 'refractive adaptation' and 'occlusion.' Our aim is to provide guidelines for patient management based, for the first time, on experimentally determined and statistically verifiable relationships between treatment and outcome.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 8 years of age;
* Presence of anisometropia and/or strabismus;
* inter-ocular acuity difference of at least 0.1 logMAR
* parental consent

Exclusion Criteria:

* history of previous occlusion therapy
* ocular pathology
* learning difficulties

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100
Dates: Start 2002-02; Study Completion 2005-05

PRIMARY OUTCOMES:
The primary outcome measure was logMAR visual acuity, measured 6-weekly for 18 weeks in refractive adaptation phase. In occlusion phase measured 2-weekly until no further gains

CONTACTS AND LOCATIONS:
Overall Officials: Merrick J Moseley, PhD, Principal Investigator — City, University of London
Locations (2):
- United Kingdom (2):
  - St Marys Hospitals, London, Greater London
  - Hillingdon Hospital, London, Middlesex

REFERENCES:
- [Background] Moseley MJ, Stewart CE, Fielder AR, Stephens DA; MOTAS cooperative. Intermediate spatial frequency letter contrast sensitivity: its relation to visual resolution before and during amblyopia treatment. Ophthalmic Physiol Opt. 2006 Jan;26(1):1-4. doi: 10.1111/j.1475-1313.2005.00343.x. PMID 16390475
- [Background] Stewart CE, Fielder AR, Stephens DA, Moseley MJ. Treatment of unilateral amblyopia: factors influencing visual outcome. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3152-60. doi: 10.1167/iovs.05-0357. PMID 16123414
- [Background] Stewart CE, Moseley MJ, Fielder AR, Stephens DA; MOTAS Cooperative. Refractive adaptation in amblyopia: quantification of effect and implications for practice. Br J Ophthalmol. 2004 Dec;88(12):1552-6. doi: 10.1136/bjo.2004.044214. PMID 15548811
- [Background] Stewart CE, Moseley MJ, Stephens DA, Fielder AR. Treatment dose-response in amblyopia therapy: the Monitored Occlusion Treatment of Amblyopia Study (MOTAS). Invest Ophthalmol Vis Sci. 2004 Sep;45(9):3048-54. doi: 10.1167/iovs.04-0250. PMID 15326120
- [Background] Stewart CE, Fielder AR, Stephens DA, Moseley MJ. Design of the Monitored Occlusion Treatment of Amblyopia Study (MOTAS). Br J Ophthalmol. 2002 Aug;86(8):915-9. doi: 10.1136/bjo.86.8.915. PMID 12140215
- [Background] Stewart CE, Moseley MJ, Fielder AR. Defining and measuring treatment outcome in unilateral amblyopia. Br J Ophthalmol. 2003 Oct;87(10):1229-31. doi: 10.1136/bjo.87.10.1229. PMID 14507754
- [Derived] Wallace MP, Stewart CE, Moseley MJ, Stephens DA, Fielder AR; Monitored Occlusion Treatment Amblyopia Study (MOTAS) Cooperatives; Randomized Occlusion Treatment Amblyopia Study (ROTAS) Cooperatives. Compliance with occlusion therapy for childhood amblyopia. Invest Ophthalmol Vis Sci. 2013 Sep 17;54(9):6158-66. doi: 10.1167/iovs.13-11861. PMID 23882695
- [Derived] Stewart CE, Stephens DA, Fielder AR, Moseley MJ; ROTAS Cooperative. Objectively monitored patching regimens for treatment of amblyopia: randomised trial. BMJ. 2007 Oct 6;335(7622):707. doi: 10.1136/bmj.39301.460150.55. Epub 2007 Sep 13. PMID 17855283